CLINICAL TRIAL: NCT02988921
Title: MRI and CT Simulation in the Evaluation of Tumor Response and Target Volume Definition for Esophageal or Esophagogastric Cancer Patients Undergoing Chemoradiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XIN WANG, MD, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-161/1240
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Esophagus Cancer; Esophagogastric Junction Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel

ARMS (1):
- Esophageal or esophagogastric cancer (Experimental)
  Interventions: Device: MRI and CT; Radiation: Ratiotherapy; Drug: Paclitaxel, platinum-based drug

INTERVENTIONS:
Device: MRI and CT
Radiation: Ratiotherapy
Drug: Paclitaxel, platinum-based drug

SUMMARY:
Magnetic resonance imaging (MRI) with functional features of diffusion weighted imaging (DWI) are advancing imaging technologies that have potential to overcome limitations of conventional staging methods, radiation treatment planning and the assessment of tumor response in esophageal or esophagogastric cancer. This study aimed to explore the value of MRI for the prediction of tumor response to chemoradiotherapy and accurate target volume delineation as compared to CT simulation for patients with unresectable or potentially resectable esophageal or esophagogastric cancer undergoing chemoradiotherapy. The average CT texture features are also extracted before and during treatment to establish a model to predict the prognosis or side effects (e.g. radiation pneumonitis or esophagitis) of patients.

DETAILED DESCRIPTION:
1. Both DW-MRI and CT simulation will be performed before chemoradiotherapy and after 18-22 fractions. Also MRI will be performed after treatment. The investigators will contour based on the MRI image and compare this with the standard CT plan before and during treatment.
2. The predictive potential of initial tumor ADC, and change in ADC during and after treatment for tumor response will be assessed.
3. The average CT texture features not only in the present study but also of those who treated previously in our department (since 2014) will be extracted before and during chemoradiotherapy to establish a model to predict the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma of the esophageal or esophagogastric junction
* Unresectable or potentially resectable tumor (cT3-4N0-1M0-M1a, according to AJCC 6th) based on standard primary staging by EUS and CT
* Age>18 years
* No distant metastasis other than supraclavicular lymph nodes
* No prior history of thoracic radiation or chemotherapy
* Patients must have normal organ and marrow function as defined below: Leukocytes: greater than or equal to 3,500 G/L; Platelets: greater than or equal to 100,000/mm3 .Hemoglobin:greater than or equal to 10g/L .Total bilirubin: within normal institutional limits; AST/ALT: less than or equal to 1.5 times the upper limit; Creatinine within normal upper limits
* Informed consent

Exclusion Criteria:

* Contraindication for MRI scanning
* Patients with other cancer history except cervical carcinoma in situ and non-malignant melanoma skin cancer
* Pregnant or lactating females
* Contraindication for radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response based on MRI and CT simulation | up to 8 weeks
Radiotherapy target volume assessment with pre- and post-chemoradiotherapy based on MRI and CT simulation | up to 8 weeks
Evaluation of tumor heterogeneity with IBEX software | up to 8 weeks
  Using the average CT images for texture extraction. Histogram, gradient, cooccurrence, gray-tone difference, and filtration-based techniques are used for texture feature extraction. Models incorporating texture features are established to compare to models incorporating clinical prognostic factors alone.

SECONDARY OUTCOMES:
Overall survival | 1 year
Progress free survival | 1 year
Reduction in acute and late side effects based on modified RT treatment volumes with pre- and post-chemoradiotherapy based on MRI and CT simulation | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, National Cancer Center, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China